CLINICAL TRIAL: NCT01375686
Title: Noninvasive Screening for Early Evidence of Diabetes With SCOUT DS
Acronym: NSEEDS
Status: Completed | Type: Observational
Sponsor: VeraLight, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VL-2715
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum will be stored to later analyze lipids and insulin. This will be useful in understanding metabolic disorders experienced by the patients measured. These measurements can be used directly, or combined in a manner similar to the McAuley index to understand the risk of insulin insensitivity.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Those at Risk for Type 2 diabetes: All subjects will be at risk for diabetes based on the American Diabetes Association (ADA) Standard of Care Guidelines.

SUMMARY:
The study will complete up to 500 subjects across 9 clinical sites to evaluate the precision and accuracy of SCOUT DS (Diabetes Screening) subjects at risk for type 2 diabetes. The study will involve up to two unique Scout devices at each clinical site. Each site will initially contain only a CS-1 (Commercial SCOUT 1) "A" for collection of data. As they become available, CS-1 "B"s operating with latest version of SCOUT software will be shipped to each site.

The NSEEDS study will enroll patients at-risk for type 2 diabetes who meet the study inclusion criteria (and do not meet one or more of the exclusion criteria) at approximately 9 clinical sites distributed across the United States. Eligible subjects must be at least 18 years old, not have an existing diagnosis of diabetes and, if less than 45 years old, must have a body mass index (BMI) ≥ 25 and at least one other risk factor for type 2 diabetes.

The data will be collected and a partial area under the receiver operator curve (pAUC) will be computed via the method of moments between the 20% and 50% false positive rates based on the first valid Scout "A" measurement for each patient. The impaired glucose tolerance status will be determined by the average of the two hour, post challenge plasma glucose samples measured at the central laboratory. This will be compared to 1000 bootstrap re-samplings of the calibration data pulling a cohort that matches that collected during this study. A test will be conducted to assure that the SCOUT performance lies within a 95% empirical confidence interval based on the bootstrap re-sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 45 years;

   OR
2. Age 18 to 44 years and a BMI > 25 with one or more of the following diabetes risk factors:

   * Habitually physically inactive (less than 30 minutes of moderate physical activity most, if not all, days of the week)
   * Has a first-degree relative with type 2 diabetes
   * African American, Latino, Native American, Asian American, Pacific Islander
   * Has delivered a baby weighing > 9 lb or previously diagnosed with gestational diabetes
   * Hypertension (≥140/≥ 90 mmHg) or being treated for hypertension
   * HDL cholesterol level < 35 mg/dL and/or a fasting triglyceride level ≥ 250 mg/dL or being treated for dyslipidemia with medication
   * Has been previously diagnosed with Polycystic Ovary Syndrome (PCOS)
   * Had impaired glucose tolerance or impaired fasting glucose on previous testing within the last 3 years
   * Conditions associated with insulin resistance such as severe obesity or acanthosis nigricans
   * History of vascular disease including heart attack, stroke, angina, coronary heart disease, atherosclerosis, congestive heart failure or peripheral arterial disease

Exclusion Criteria:

* Prior participation in VeraLight studies: VL-2701, VL-2710, VL-2711, VL-2712 , or VL-2718
* Diagnosed with any type of diabetes, including type 1 or 2
* Known to have, or at risk for, photosensitivity reactions ( e.g., sensitive to ultraviolet light, or taking medication known to cause photosensitivity)
* Receiving any investigational treatment in the past 14 days
* Psychosocial issues that interfere with an ability to follow study procedures
* Conditions that cause secondary diabetes including Cushing's syndrome, acromegaly, hemochromatosis, pancreatitis, or cystic fibrosis
* Taking glucose lowering medications*
* Known to be pregnant (self reported)
* Receiving dialysis or having known renal compromise
* Scars, tattoos, rashes or other disruption/discoloration on the left volar forearm.
* Recent (within past month) or current oral steroid therapy or topical steroids applied to the left forearm; inhaled steroid therapy is not excluded
* Current chemotherapy, or chemotherapy within the past 12 months
* Receiving medications that fluoresce *
* Prior bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the study, volunteers age 18 and above, of either sex and of any ethnic background, will be recruited at up to 9 clinical sites. The number of sites may be decreased as the sponsor has the right to close a site due to protocol compliance or enrollment issues during the course of the study. All subjects will be at risk for diabetes based on the American Diabetes Association Standard of Care Guidelines. Subjects in the 18-44 age range must have a BMI > 25 plus an additional risk factor for type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Validation of SCOUT DS algorithm, ROC performance equivalent to FPG, A1c for detection abnormal glucose tolerance. | 6 months
  The data will be collected and a partial area under the receiver operator curve (pAUC) will be computed via the method of moments between the 20% and 50% false positive rates based on the first valid Scout "A" measurement for each patient. The impaired glucose tolerance status will be determined by the average of the two hour, post challenge plasma glucose samples measured at the central laboratory. A test will be conducted to assure that the SCOUT performance lies within a 95% empirical confidence interval based on the bootstrap re-sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kyle, MD, Principal Investigator — Radiant Chicago; Tami Helmer, MD, Principal Investigator — Radiant Minneapolis; Michael Noss, MD, Principal Investigator — Radiant Cincinnati; William Jennings, MD, Principal Investigator — Radiant San Antonio; Daniel Brune, MD, Principal Investigator — Accelovance Peoria; Martin L Kabongo, MD, Principal Investigator — Accelovance San Diego; Earl Martin, MD, Principal Investigator — DM Clinical; Audrey Lacour, MD, Principal Investigator — JUNO Research; David Bolshoun, MD, Principal Investigator — Radiant Denver
Locations (1):
- Radiant Denver, Denver, Colorado, United States